CLINICAL TRIAL: NCT04389710
Title: Convalescent Plasma for the Treatment of Patients With COVID-19
Brief Title: Convalescent Plasma for the Treatment of COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20D.379
Record Dates: First submitted 2020-04-27; First posted 2020-05-15 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Provide access to COVID-19 convalescent plasma for patients infected with SARS-CoV-2 currently hospitalized in acute care facilities
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention Group (Experimental): Participants included in the experimental group will receive 200-600 milliliters of convalescent plasma, administered at a rate of 100-250 mL/hr
  Interventions: Drug: Convalescent Plasma

INTERVENTIONS:
Drug: Convalescent Plasma — One to two units (200-600 mL) of ABO compatible COVID-19 convalescent plasma

SUMMARY:
This protocol provides access to investigational convalescent plasma for patients in acute care facilities infected with SARS-CoV-2 who have severe or life-threatening COVID-19, or who are judged by a healthcare provider to be at high risk of progression to severe or life-threatening disease. Following provision of informed consent, patients will be transfused with 1-2 units of ABO compatible convalescent plasma obtained from an individual who has recovered from documented infection with SARS-CoV-2 (as detailed in separate protocol). Safety information collected will include serious adverse events judged to be related to administration of convalescent plasma. Other information to be collected will include patient demographics, acute care facility resource utilization (total length of stay, days in ICU, days intubated), and survival to discharge from acute care facility.

DETAILED DESCRIPTION:
This is an open-label expanded access program to make appropriately matched convalescent plasma available for the treatment of patients in acute care facilities infected with SARS-CoV-2 who have severe or life-threatening COVID-19, or who are judged by a healthcare provider to be at high risk of progression to severe or life-threatening disease. COVID-19 convalescent plasma will be obtained from the Jefferson Blood Bank and will meet all regulatory requirements for conventional plasma and FDA's additional considerations for COVID-19 convalescent plasma (https://www.fda.gov/vaccines-blood-biologics/investigational-new-drug-ind-or-device-exemption-ide-process-cber/investigational-covid-19-convalescent-plasma-emergency-inds).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Laboratory confirmed diagnosis of SARS-CoV-2
* Admitted to an acute care facility for the treatment of COVID-19 complications
* Informed consent provided by patient or legally authorized representative
* Severe or life threatening COVID-19, or judged by the treating provider to be at high risk of progression to severe or life-threatening disease

Severe Disease defined as any of the following

* Dyspnea
* Respiratory rate > 30/minute
* Oxygen saturation <94%
* Partial pressure of arterial oxygen to fraction of inspired oxygen ratio <300
* Lung infiltrates >50% within 24 to 48 hours

Life-threatening disease defined as any of the following

* Respiratory failure
* Septic shock
* Multiple organ dysfunction or failure • Informed consent provided by patient or healthcare proxy

Exclusion Criteria:

* Receipt of pooled immunoglobulin in past 30 days
* Contraindication to transfusion or history of prior reactions to transfusion blood products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
Number of patients who receive COVID-19 convalescent plasma transfusions in acute care facilities infected with SARS-CoV-2 | 1 year
  Number of patients who are consented and ultimately receive convalescent plasma transfusion.

SECONDARY OUTCOMES:
Number and type of adverse events associated with COVID-19 convalescent plasma in patients with COVID-19 | 0, 1, 2, 3, 7, 14 days
  Adverse Events including transfusion reaction (fever, rash), transfusion related acute lung injury (TRALI), transfusion associated circulatory overload (TACO), and transfusion infection
Length of hospital stay | 0, 1, 2, 3, 7, 14, 28, 60, and 90 days
  Days of hospitalization
Length of Intensive Care Unit stay | 0, 1, 2, 3, 7, 14, 28, 60, and 90 days
  Days of Intensive Care Unit management
Length of intubation | 0, 1, 2, 3, 7, 14, 28, 60, and 90 days
  Days of intubation requirement
Survival to discharge | 0, 1, 2, 3, 7, 14, 28, 60, and 90 days
  Proportion of patients who are successfully discharged from acute care facility
Changes in complete blood count in patients after receiving convalescent plasma | 0 and 7 days
  Laboratory values will be evaluated at day 0 and 7 (or the day of hospital discharge, if sooner).
Abnormal changes in Basic Metabolic Panel (BMP) measures in patients after receiving convalescent plasma | 0 and 7 days
  BMP tests include measures of glucose, calcium, sodium, potassium, bicarbonate, chloride, blood urea nitrogen, and creatinine. Changes of interest include those that are flagged as abnormal. Laboratory values will be evaluated at day 0 and 7 (or the day of hospital discharge, if sooner).
Changes in C-Reactive Protein (CRP) in patients after receiving convalescent plasma | 0 and 7 days
  Laboratory values will be evaluated at day 0 and 7 (or the day of hospital discharge, if sooner).
Changes in d-dimer in patients after receiving convalescent plasma | 0 and 7 days
  Laboratory values will be evaluated at day 0 and 7 (or the day of hospital discharge, if sooner).
Changes in fibrinogen in patients after receiving convalescent plasma | 0 and 7 days
  Laboratory values will be evaluated at day 0 and 7 (or the day of hospital discharge, if sooner).
Changes in prothrombin time (PT) in patients after receiving convalescent plasma | 0 and 7 days
  Laboratory values will be evaluated at day 0 and 7 (or the day of hospital discharge, if sooner).
Changes in partial thromboplastin time (PTT) in patients after receiving convalescent plasma | 0 and 7 days
  Laboratory values will be evaluated at day 0 and 7 (or the day of hospital discharge, if sooner).

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States